CLINICAL TRIAL: NCT05566665
Title: Nosocomial Infections in Patients Treated With Extracorporeal Membrane Oxygenation
Brief Title: Nosocomial Infections in ECMO Patients
Acronym: INF-ECMO
Status: Recruiting | Type: Observational
Sponsor: Policlinico Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Giacomo Grasselli, Full Professor of Anesthesiology and Intensive Care Medicine, Director of General Intensive Care Unit, Principal Investigator, Policlinico Hospital
Other Study IDs: INF-ECMO
Record Dates: First submitted 2022-09-13; First posted 2022-10-04 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Acute Respiratory Distress Syndrome; Nosocomial Infection; Extracorporeal Membrane Oxygenation Complication
MeSH Terms: conditions — Respiratory Distress Syndrome; Cross Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and bronchoalveolar lavage (BAL) samples will be collected. Blood samples collection timepoint: just prior to administration of the fifth dose of antibiotic (i.e., after 48 hours of therapy) (t0); at 1 hour after the end of the infusion (t1); 2 hours after the infusion (t2); 4 hours after the infusion (t3). They will be centrifuged, and plasma samples stored at -20°c until analysis. BAL samples will be collected only at t0. BAL will be carried out following standard procedure. The sample will be fresh-frozen and cryopreserved at -80°C. Cryopreserved samples will be shipped to the collaborating center (ASST Fatebenefratelli Sacco, Milan, Italy) at the end of the recruitment period, and thus tests will be performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ECMO requiring ARDS patients: The study population for the Aim 1 study will comprise adult patients admitted to the participating ICUs suffering from ARDS (as defined by the Berlin criteria) and treated with ECMO.
  The study population for the Aim 2 study will comprise the subgroup of patients as per Aim 1, whose clinical course is complicated by VAP necessitating antibiotic treatment with ceftazidime/avibactam, meropenem/vaborbactam, ceftolozane/tazobactam, or cefiderocol.
- Antibiotic treated ECMO requiring ARDS patients.: The study population for the Aim 2 study will comprise the subgroup of patients as per Aim 1, whose clinical course is complicated by VAP necessitating antibiotic treatment with ceftazidime/avibactam, meropenem/vaborbactam, ceftolozane/tazobactam, or cefiderocol.
  Interventions: Diagnostic Test: Collection of blood and bronchoalveolar samples to study Pharmacokinetics of ceftazidime/avibactam, meropenem/varbobactam, ceftolozane/tazobactam, or cefiderocol

INTERVENTIONS:
Diagnostic Test: Collection of blood and bronchoalveolar samples to study Pharmacokinetics of ceftazidime/avibactam, meropenem/varbobactam, ceftolozane/tazobactam, or cefiderocol — The antibiotic treatment with ceftazidime/avibactam, meropenem/vaborbactam, ceftolozane/tazobactam, or cefiderocol will follow the standard clinical practice.
  The concentration of ceftazidime/avibactam, meropenem/vaborbactam, ceftolozane/tazobactam, or cefiderocol will be measured at specific timepoints in plasma samples and bronchoalveolar lavage samples, and a PK analysis and modeling will be carried out .
  Groups: Antibiotic treated ECMO requiring ARDS patients.

SUMMARY:
Nosocomial Infections (NI) are a common and dreadful complication for patients suffering from Acute Respiratory Distress Syndrome (ARDS) treated with Extracorporeal Membrane Oxygenation (ECMO). Unfortunately, no study has thoroughly evaluated NI in this fragile patient cohort. Newly developed antibiotics may help manage such infections, but their pharmacokinetics (PK) during ECMO has not been evaluated.

Objectives of this prospective observational multicenter pharmacological no-profit study are: 1) describe incidence, microbial etiology, and resistance patterns, and assess risk factors for NIs in a large prospective cohort of ARDS patients undergoing ECMO. 2) provide a PK analysis of ceftazidime/avibactam, meropenem/vaborbactam, ceftolozane/tazobactam, and cefiderocol in adult patients undergoing ECMO Incidence, microbial etiology, and antibiotic resistance patterns of confirmed NIs will be prospectively collected and analyzed. In the subgroup of patients treated with ceftazidime/avibactam, meropenem/vaborbactam, ceftolozane/tazobactam, or cefiderocol as per clinical practice, blood and bronchoalveolar concentration of the antibiotic will be measured, and PK modeling carried out.

DETAILED DESCRIPTION:
The most severe acute respiratory distress syndrome (ARDS) cases require extracorporeal membrane oxygenation (ECMO). ECMO is a life-support technique utilized in patients with reversible refractory respiratory failure. Nosocomial infections (NI) are common complications in ECMO patients due to predisposing factors such as patients' comorbidities, immunocompromise associated with the critical illness, and invasiveness of ECMO and other life support procedures. Few studies have assessed the incidence, risk factors, microbial etiology, and antibiotic resistance of NIs during ECMO. In a monocentric retrospective observational analysis, a high incidence of NI was detected in ECMO patients. The most common NI was ventilation-associated pneumonia (VAP), frequently caused by multidrug-resistant (MDR) bacteria. Patients developing an infection had a longer duration of ECMO and mechanical ventilation and a more prolonged ICU stay. The rate of MDR bacterial isolates was very high, and the first NI episode caused by MDR germs was an independent risk factor for death. To date, no prospective study has studied the epidemiology and clinical significance of NIs during ECMO. Better knowledge of NIs epidemiology during ECMO may allow us to target possibly causative agents using more specific empirical antibiotic therapy, increase accuracy, and optimize the timing of antimicrobial treatment. In turn, this may lead to better treatment of NIs in patients undergoing ECMO, thus reducing the overall burden of infections in such a fragile population and allowing a significant decrease in the costs of treatment.

Several new antimicrobial agents utilized for the treatment of MDR infections (i.e., ceftazidime/avibactam, meropenem/vaborbactam, ceftolozane/tazobactam, cefiderocol) have been granted approval in Europe for the treatment of VAP. Antibiotic efficacy in pneumonia requires sufficient unbound drug concentrations at the pulmonary site of infection, and determination of the bronchopulmonary availability of antibiotics in epithelial lining fluid (ELF) allows penetration into the lung to be characterized. While population pharmacokinetic (PK) models have been carried out in healthy volunteers, no data is available relative to the PK of those antibiotics ECMO patients. In general, ECMO has been shown to impact PK in three primary ways: direct extraction by the circuit increased volume of distribution, and altered clearance5. Thus, knowledge of the PK of these newly introduced antibiotic agents in ECMO patients suffering from VAP due to MDR bacteria may be of great clinical impact.

Based on these premises, in a large cohort of ECMO patients with ARDS, the investigators will carry out a prospective multicenter observational study to describe NIs and their risk factors. Overall, with this study, the investigators will significantly broaden the data as regards to NIs during ECMO.

In addition, in a subgroup of patients treated with ceftazidime/avibactam, meropenem/vaborbactam, ceftolozane/tazobactam, or cefiderocol for VAP during ECMO treatment, the investigators will carry out a pharmacokinetic study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of ARDS (i.e., acute onset ( < 7 days) from the known clinical insult of respiratory failure, with bilateral opacities - not explained by effusions, lung and lobar collapse, or nodules -, not fully explained by cardiac failure/fluid overload; with P/F ratio <= 300 mmHg and continuous positive airway pressure >= 5 cmH2O)
* Ongoing ECMO

Adjunctive Inclusion Criterium for the sole Secondary Objective:

- Antibiotic treatment with ceftazidime/avibactam, meropenem/vaborbactam, ceftolozane/tazobactam, or cefiderocol.

Exclusion Criteria:

* Pregnancy
* Expected survival < 24 hours.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for the Aim 1 study will comprise adult patients admitted to the aforementioned ICUs suffering from ARDS (as defined by the Berlin criteria) and treated with ECMO.
  The study population for the Aim 2 study will comprise the subgroup of patients as per Aim 1, whose clinical course is complicated by VAP necessitating antibiotic treatment with ceftazidime/avibactam, meropenem/vaborbactam, ceftolozane/tazobactam, or cefiderocol
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of NIs in a large prospective cohort of ARDS patients undergoing ECMO. | January 2023-December 2024
  Only microbiologically-confirmed infections will be considered. Accordingly, the composite outcome (i.e., infected patient) will be composed of the following NIs: ventilator-associated pneumonia (VAP), catheter-associated urinary tract infection (UTI), bloodstream infection (BSI), and catheter-related bloodstream infection (CRBSI). Incidence of pulmonary aspergillosis and clostridium difficile colitis will be collected but not included in the composite outcome (i.e., infected patient). To carry out this aim, a supervisor for each participating center will be in charge of patients' follow-up. For each center, a critical care specialist and an infectious disease specialist will review the available clinical and laboratory data. Incidence will be expressed as: 1) percentage of patients who will develop a NI/total of patients; 2) rate of incidence: number of infection/total time at risk of NIs.
Microbial etiology of NIs in a large prospective cohort of ARDS patients undergoing ECMO. | January 2023-December 2024
  Only microbiologically-confirmed infections will be considered. Accordingly, the composite outcome (i.e., infected patient) will be composed of the following NIs: ventilator-associated pneumonia (VAP), catheter-associated urinary tract infection (UTI), bloodstream infection (BSI), and catheter-related bloodstream infection (CRBSI). Incidence of pulmonary aspergillosis and clostridium difficile colitis will be collected but not included in the composite outcome (i.e., infected patient). To carry out this aim, a supervisor for each participating center will be in charge of patients' follow-up. For each center, a critical care specialist and an infectious disease specialist will review the available clinical and laboratory data. Different microbial etiology will be described according to simple descriptive statistics methods.
Resistance patterns of NIs in a large prospective cohort of ARDS patients undergoing ECMO. | January 2023-December 2024
  Only microbiologically-confirmed infections will be considered. Accordingly, the composite outcome (i.e., infected patient) will be composed of the following NIs: ventilator-associated pneumonia (VAP), catheter-associated urinary tract infection (UTI), bloodstream infection (BSI), and catheter-related bloodstream infection (CRBSI). Incidence of pulmonary aspergillosis and clostridium difficile colitis will be collected but not included in the composite outcome (i.e., infected patient). To carry out this aim, a supervisor for each participating center will be in charge of patients' follow-up. For each center, a critical care specialist and an infectious disease specialist will review the available clinical and laboratory data. Resistance patterns of NIs' microbes will be described according to simple descriptive statistics methods.
Risk factors of NIs in a large prospective cohort of ARDS patients undergoing ECMO. | January 2023-December 2024
  Only microbiologically-confirmed infections will be considered. Accordingly, the composite outcome (i.e., infected patient) will be composed of the following NIs: ventilator-associated pneumonia (VAP), catheter-associated urinary tract infection (UTI), bloodstream infection (BSI), and catheter-related bloodstream infection (CRBSI). Incidence of pulmonary aspergillosis and clostridium difficile colitis will be collected but not included in the composite outcome (i.e., infected patient). To carry out this aim, a supervisor for each participating center will be in charge of patients' follow-up. For each center, a critical care specialist and an infectious disease specialist will review the available clinical and laboratory data. Multivariate analysis will be conducted to evaluate risk factors of NIs. For each risk factor identified Odds Ratio with 95% Confidence Interval will be reported.

SECONDARY OUTCOMES:
Plasma concentration of ceftazidime/avibactam, meropenem/vaborbactam, ceftolozane/tazobactam, and cefiderocol in adult patients undergoing ECMO | January 2023-December 2024
  For this aim, there will be no modification of patients' treatment and antibiotic use. The antibiotic treatment with ceftazidime/avibactam, meropenem/vaborbactam, ceftolozane/tazobactam, or cefiderocol will follow the standard clinical practice.
  The concentration of ceftazidime/avibactam, meropenem/vaborbactam, ceftolozane/tazobactam, or cefiderocol will be measured in plasma samples at four specific timepoints (the first before the 5th administration of antibiotic, and then 1, 2 and 4 hours after the administration) to evaluate Maximum Plasmatic Concentration of antibiotic and its pharmacokinetics.
Bronchoalveolar lavage concentration of ceftazidime/avibactam, meropenem/vaborbactam, ceftolozane/tazobactam, and cefiderocol in adult patients undergoing ECMO | January 2023-December 2024
  For this aim, there will be no modification of patients' treatment and antibiotic use. The antibiotic treatment with ceftazidime/avibactam, meropenem/vaborbactam, ceftolozane/tazobactam, or cefiderocol will follow the standard clinical practice.
  The concentration of ceftazidime/avibactam, meropenem/vaborbactam, ceftolozane/tazobactam, or cefiderocol will be measured in bronchoalveolar lavage (BAL) samples before the 5th administration of antibiotic to evaluate BAL Concentration of antibiotic.

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Scaravilli, MD, Principal Investigator — University of Milan; Giacomo Grasselli, MD, Principal Investigator — University of Milan
Locations (2):
- Italy (2):
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, MI
  - Fondazione IRCCS Ca'Granda - Ospedale Maggiore Policlinico, Milan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available online already
Access Criteria: Open access
URL: http://INFECMO.unimi.it

REFERENCES:
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Schmidt M, Hajage D, Lebreton G, Monsel A, Voiriot G, Levy D, Baron E, Beurton A, Chommeloux J, Meng P, Nemlaghi S, Bay P, Leprince P, Demoule A, Guidet B, Constantin JM, Fartoukh M, Dres M, Combes A; Groupe de Recherche Clinique en REanimation et Soins intensifs du Patient en Insuffisance Respiratoire aiguE (GRC-RESPIRE) Sorbonne Universite; Paris-Sorbonne ECMO-COVID investigators. Extracorporeal membrane oxygenation for severe acute respiratory distress syndrome associated with COVID-19: a retrospective cohort study. Lancet Respir Med. 2020 Nov;8(11):1121-1131. doi: 10.1016/S2213-2600(20)30328-3. Epub 2020 Aug 13. PMID 32798468
- [Background] Grasselli G, Scaravilli V, Di Bella S, Biffi S, Bombino M, Patroniti N, Bisi L, Peri AM, Pesenti A, Gori A, Alagna L. Nosocomial Infections During Extracorporeal Membrane Oxygenation: Incidence, Etiology, and Impact on Patients' Outcome. Crit Care Med. 2017 Oct;45(10):1726-1733. doi: 10.1097/CCM.0000000000002652. PMID 28777198
- [Background] Yusuf E, Bax HI, Verkaik NJ, van Westreenen M. An Update on Eight "New" Antibiotics against Multidrug-Resistant Gram-Negative Bacteria. J Clin Med. 2021 Mar 4;10(5):1068. doi: 10.3390/jcm10051068. PMID 33806604
- [Background] Sherwin J, Heath T, Watt K. Pharmacokinetics and Dosing of Anti-infective Drugs in Patients on Extracorporeal Membrane Oxygenation: A Review of the Current Literature. Clin Ther. 2016 Sep;38(9):1976-94. doi: 10.1016/j.clinthera.2016.07.169. Epub 2016 Aug 21. PMID 27553752
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Falcone M, Menichetti F, Cattaneo D, Tiseo G, Baldelli S, Galfo V, Leonildi A, Tagliaferri E, Di Paolo A, Pai MP. Pragmatic options for dose optimization of ceftazidime/avibactam with aztreonam in complex patients. J Antimicrob Chemother. 2021 Mar 12;76(4):1025-1031. doi: 10.1093/jac/dkaa549. PMID 33378458
- [Background] Castagnola E, Cangemi G, Mesini A, Castellani C, Martelli A, Cattaneo D, Mattioli F. Pharmacokinetics and pharmacodynamics of antibiotics in cystic fibrosis: a narrative review. Int J Antimicrob Agents. 2021 Sep;58(3):106381. doi: 10.1016/j.ijantimicag.2021.106381. Epub 2021 Jun 19. PMID 34157401
- [Background] Grasselli G, Scaravilli V, Mangioni D, Scudeller L, Alagna L, Bartoletti M, Bellani G, Biagioni E, Bonfanti P, Bottino N, Coloretti I, Cutuli SL, De Pascale G, Ferlicca D, Fior G, Forastieri A, Franzetti M, Greco M, Guzzardella A, Linguadoca S, Meschiari M, Messina A, Monti G, Morelli P, Muscatello A, Redaelli S, Stefanini F, Tonetti T, Antonelli M, Cecconi M, Foti G, Fumagalli R, Girardis M, Ranieri M, Viale P, Raviglione M, Pesenti A, Gori A, Bandera A. Hospital-Acquired Infections in Critically Ill Patients With COVID-19. Chest. 2021 Aug;160(2):454-465. doi: 10.1016/j.chest.2021.04.002. Epub 2021 Apr 20. PMID 33857475